CLINICAL TRIAL: NCT03404726
Title: An Open-label, Multicenter Phase 1 Study to Characterize the Safety, Tolerability, Preliminary Antileukemic Activity, Pharmacokinetics, and Maximum Tolerated Dose or Pharmacological Active Dose of BAY2402234 in Patients With Advanced Myeloid Malignancies
Brief Title: A Study to Investigate BAY2402234, a Dihydroorotate Dehydrogenase (DHODH) Inhibitor, in Myeloid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of sufficient clinical benefit
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19420; 2017-002896-24 (EudraCT Number)
Record Dates: First submitted 2017-11-29; First posted 2018-01-19 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Leukemia
Keywords: Acute myeloid leukemia; Myelodysplastic Syndromes; Chronic myelomonocytic leukemia; Dihydroorotate dehydrogenase (DHODH) inhibitor
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — orludodstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Dose escalation with sequential cohorts enrolling patients with AML, MDS, or CMML. Patients will be treated in 28-day cycles with once daily oral administration of BAY2402234
  Interventions: Drug: BAY2402234
- Dose Expansion: AML (Experimental): After completion of dose escalation, an expansion cohort comprised of patients with AML will start. These patients will be treated in 28 day cycles with once daily oral administration of BAY2402234 at the maximum tolerated dose or pharmacologically active dose.
  Interventions: Drug: BAY2402234
- Dose Expansion: MDS (Experimental): After completion of dose escalation, an expansion cohort comprised of patients with MDS will start. These patients will be treated in 28 day cycles with once daily oral administration of BAY2402234 at the maximum tolerated dose or pharmacologically active dose.
  Interventions: Drug: BAY2402234

INTERVENTIONS:
Drug: BAY2402234 — BAY2402234 is a potent and selective small molecule inhibitor of dihydroorotate dehydrogenase. A solution of BAY2402234 will be available to initiate the trial and there are plans to transition to a tablet form of BAY2402234 once it becomes available. Both liquid and tablet formulations of BAY2402234 will be continually administered once daily by mouth in 28 day cycles.

SUMMARY:
The primary objective is to determine the safety, tolerability, pharmacokinetics, maximum tolerated dose (MTD), or pharmacological active dose (PAD) of BAY2402234 in patients with acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or chronic myelomonocytic leukemia (CMML).

The secondary objective is to evaluate evidence of clinical efficacy associated with BAY2402234 in patients with AML (defined as Complete remission, Complete remission with partial hematologic recovery), and MDS (defined as hematological improvement).

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory AML. Relapsed AML is defined as relapse after achieving a response to initial therapy and refractory AML is defined as failure to achieve a response after one previous line of therapy. Response is defined as per IWG criteria (CR, CRi or CRp). Patients who are not candidates to receive or who decline standard of care therapy are also eligible.
* Patients with intermediate-1 or higher risk MDS who have failed therapy with a hypomethylating agent, or have failed lenalidomide therapy if harboring a 5q-chromosomal deletion.
* Patients with relapsed/refractory CMML.
* Estimated glomerular filtration rate (eGFR) > 40 mL per 1.73 m^2
* Patients must have adequate coagulation (international normalized ratio [INR] ≤ 1.5; activated partial thromboplastin time [aPTT] ≤1.5 X the upper limit of normal [ULN]; patients on chronic anticoagulation therapy at investigator's discretion; patients on chronic use of direct-acting oral anticoagulants who have acceptable benefit-risk ratio at investigator's discretion)
* Adequate liver function (total bilirubin ≤1.5 X ULN (or ≤3 X ULN in patients with documented Gilbert's syndrome or for patients with hyperbilirubinemia considered due to myeloid disease), alanine aminotransferase [ALT] and aspartate aminotransferase [AST] ≤3 X ULN (or ≤5 X ULN for patients with liver involvement of their myeloid disease)

Exclusion Criteria:

* Patients eligible for hematopoietic stem cell transplantation
* Clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia
* Human immunodeficiency virus (HIV) infection
* Chronic or active hepatitis B or C if not controlled by antiviral therapy
* History of organ allograft (allogeneic bone marrow or stem cell transplant) within 3 months prior to first dose of study drug
* Serious, uncontrolled infection requiring systemic antibiotic, antifungal or antiviral therapy. Prophylactic antibiotic, antifungal and/or antiviral therapy is permitted
* Left ventricular ejection fraction (LVEF) <40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 42 days after the first dose
  The MTD was defined as the maximum dose administered during Cycle 1 at which the estimated dose-limiting toxicity (DLT) probability is closest to 30%.
Number of subjects with DLTs | Up to 42 days after the first dose
  A dose-limiting toxicity (DLT) was defined as any of the events that are clearly unrelated to underlying disease and occurring at any particular dose level during the first 28 days (i.e. Cycle 1) of treatment for non-hematological DLTs, or 42 days after the start of treatment, in the absence of active disease (i.e. < 5% blasts in bone marrow and absence of leukemic blasts in peripheral blood) for hematological DLTs. The National Cancer Institute Common Terminology Criteria for Adverse Events Version (CTCAE) v4.03 will be used to assess toxicities.
AUC(0-24) (area under the concentration versus time curve from time zero to 24 hours) after single dose on Cycle 1 Day 1 (C1D1) | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after dose administration at C1D1
Cmax (maximum observed drug concentration in plasma after single dose administration) on C1D1 | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours (QD cohorts=until 24 hours; BID cohort=until 12 hours) after dose administration at C1D1
AUC(0-24)md (AUC(0-24) after multiple dose) on Cycle 1 Day 15 (C1D15) | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after dose administration at C1D15
Cmax,md (Cmax after multiple dose) on C1D15 | Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours (QD cohorts=until 24 hours; BID cohort=until 12 hours) after dose administration at C1D1
Number of subjects with Treatment Emergent Adverse Events (TEAEs) | From first application of study intervention up to 30 days after end of treatment
  An AE was any untoward medical occurrence (i.e. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation subject after providing written informed consent for participation in the study.

SECONDARY OUTCOMES:
Number of acute myeloid leukemia (AML) patients with complete remission (CR) and complete response with partial recovery of peripheral blood counts (CRh) | Up to 6 months on average
Number of myelodysplastic syndrome (MDS) patients with hematologic improvement (erythroid response, platelet response, and neutrophil response) | Every month until disease progression or patient was withdrawn from study, up to 6 months on average

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/